CLINICAL TRIAL: NCT02986243
Title: Preparing for Kidney Transplant by Attaining a Healthy Weight
Acronym: FFC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-1593
Record Dates: First submitted 2016-11-30; First posted 2016-12-08 (Estimated); Last update posted 2025-02-19 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects receive a diet plan and exercise regimen.
  Interventions: Other: Exercise; Dietary Supplement: Diet Plan

INTERVENTIONS:
Other: Exercise — 6 months worth of exercise regimen
Dietary Supplement: Diet Plan — Each subject will receive a personalized diet plan from nutritionist.

SUMMARY:
The purpose of this study is to determine if an assigned physical fitness program will result in weight loss to prepare patients for kidney transplant.

DETAILED DESCRIPTION:
The goal of this study is to prepare subjects for kidney transplant. Patients who are in need of a kidney transplant but are unable to be place on the wait list due to weight will be enrolled in a six month workout program. The workout program will consist of counseling from a registered dietician, personal training from certified trainers and constant health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age and older but less than 65
* All patients who are currently listed as "inactive" on the University of Chicago kidney transplant wait list
* Those with a body mass index of 40-44
* Those with access to the Internet
* Have transportation to the fitness center (Formula Fitness Center at Union Station location)

Exclusion Criteria:

* Those patients who are listed "inactive" on the wait-list due to co-morbid conditions other than obesity
* Those who are unwilling to attend fitness center appointments
* Those who do not have adequate transportation to the fitness center
* Those who do not have access to the Internet
* Those who are not comfortable navigating and using the Internet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 6 months
  The difference in starting weight and ending weight six months after beginning exercise program will be measured.

IPD SHARING:
Plan to Share IPD: No